CLINICAL TRIAL: NCT04276896
Title: Phase I/II Multicenter Trial of Lentiviral Minigene Vaccine (LV-SMENP) of Covid-19 Coronavirus
Brief Title: Immunity and Safety of Covid-19 Synthetic Minigene Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Third People's Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20001
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Pathogen Infection Covid-19 Infection
Keywords: Lentiviral vector; LV-DC vaccine; Covid-19 CTL
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pathogen-specific DC and CTLs (Experimental): Patients will receive approximately 5x10^6 LV-DC vaccine and 1x10^8 CTLs via sub-cutaneous injections and iv infusions, respectively.
  Interventions: Biological: Injection and infusion of LV-SMENP-DC vaccine and antigen-specific CTLs

INTERVENTIONS:
Biological: Injection and infusion of LV-SMENP-DC vaccine and antigen-specific CTLs — Patients will receive approximately 5x10^6 LV-DC vaccine and 1x10^8 CTLs via sub-cutaneous injections and iv infusions, respectively.

SUMMARY:
In December 2019, viral pneumonia caused by a novel beta-coronavirus (Covid-19) broke out in Wuhan, China. Some patients rapidly progressed and suffered severe acute respiratory failure and died, making it imperative to develop a safe and effective vaccine to treat and prevent severe Covid-19 pneumonia. Based on detailed analysis of the viral genome and search for potential immunogenic targets, a synthetic minigene has been engineered based on conserved domains of the viral structural proteins and a polyprotein protease. The infection of Covid-19 is mediated through binding of the Spike protein to the ACEII receptor, and the viral replication depends on molecular mechanisms of all of these viral proteins. This trial proposes to develop and test innovative Covid-19 minigenes engineered based on multiple viral genes, using an efficient lentiviral vector system (NHP/TYF) to express viral proteins and immune modulatory genes to modify dendritic cells (DCs) and to activate T cells. In this study, the safety and efficacy of this LV vaccine (LV-SMENP) will be investigated.

DETAILED DESCRIPTION:
Background: The 2019 discovered new coronavirus, Covid-19, is an enveloped positive strand single strand RNA virus. The number of Covid-19 infected people has increased rapidly and WHO has warned that the spread of Covid-19 may soon become pandemic and have disastrous outcomes. Covid-19 could pose a serious threat to human health and global economy. There is no vaccine available or clinically approved antiviral therapy as yet. This study aims to evaluate the safety and efficacy of treating Covid-19 infections with a novel lentiviral based DC and T cell vaccines.

Objective: Primary study objectives: Injection and infusion of LV-SMENP DC and antigen-specific cytotoxic T cell vaccines to healthy volunteers and Covid-19 infected patients to evaluate the safety.

Secondary study objectives: To evaluate the anti- Covid-19 efficacy of the LV-SMENP DC and antigen-specific cytotoxic T cell vaccines.

Design:

1. Based on the genomic sequence of the new coronavirus Covid-19, select conserved and critical structural and protease protein domains to engineer lentiviral SMENP minigenes to express Covid-19 antigens.
2. LV-SMENP-DC vaccine is made by modifying DC with lentivirus vectors expressing Covid-19 minigene SMENP and immune modulatory genes. CTLs will be activated by LV-DC presenting Covid-19 specific antigens.
3. LV-DC vaccine and antigen-specific CTLs are prepared in 7~21 days. Subject will receive total 5x10^6 cells of LV-DC vaccine and 1x10^8 antigen-specific CTLs via sub-cutaneous injection and IV infusion, respectively. Patients are followed weekly for one month after the infusion, monthly for 3 months, and then every 3 months until the trial ends.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory (RT-PCR) confirmed Covid-19 infection in throat swab and/or sputum and/or lower respiratory tract samples;
* The interval between the onset of symptoms and randomized is within 7 days. The onset of symptoms is mainly based on fever. If there is no fever, cough or other related symptoms can be used;
* White blood cells ≥ 3,500 / μl, lymphocytes ≥ 750 / μl;
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or tuberculosis (TB) test is negative;
* Sign the Informed Consent Form on a voluntary basis;

Exclusion Criteria:

* Subject infected with HCV (HCV antibody positive), HBV (HBsAg positive), HIV (HIV antibody positive), or HTLV (HTLV antibody positive).
* Subject is albumin-intolerant.
* Subject with life expectancy less than 4 weeks.
* Subject participated in other investigational somatic cell therapies within past 30 days.
* Subject with positive pregnancy test result.
* Researchers consider unsuitable.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-24 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement based on the 7-point scale | 28 days after randomization
  A decline of 2 points on the 7-point scale from admission means better outcome. The 7-category ordinal scale that ranges from 1 (discharged with normal activity) to 7 (death).
Lower Murray lung injury score | 7 days after randomization
  Murray lung injury score decrease more than one point means better outcome. The Murray scoring system range from 0 to 4 according to the severity of the condition.

SECONDARY OUTCOMES:
28-day mortality | Measured from Day 0 through Day 28
  Number of deaths during study follow-up
Duration of mechanical ventilation | Measured from Day 0 through Day 28
  Duration of mechanical ventilation use in days. Multiple mechanical ventilation durations are summed up.
Duration of hospitalization | Measured from Day 0 through Day 28
  Days that a participant spent at the hospital. Multiple hospitalizations are summed up.
Proportion of patients with negative RT-PCR results | 7 and 14 days after randomization
  Proportion of patients with negative RT-PCR results of virus in upper and/or lower respiratory tract samples.
Proportion of patients in each category of the 7-point scale | 7,14 and 28 days after randomization
  Proportion of patients in each category of the 7-point scale, the 7-category ordinal scale that ranges from 1 (discharged with normal activity) to 7 (death).
Proportion of patients with normalized inflammation factors | 7 and 14 days after randomization
  Proportion of patients with different inflammation factors in normalization range.
Frequency of vaccine/CTL Events | Measured from Day 0 through Day 28
  Frequency of vaccine/CTL Events
Frequency of Serious vaccine/CTL Events | Measured from Day 0 through Day 28
  Frequency of Serious vaccine/CTL Events

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (3):
- China (3):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No